CLINICAL TRIAL: NCT05067192
Title: Optimization of Morphomer-based Alpha-synuclein PET Tracers
Status: Completed | Type: Observational
Sponsor: Skane University Hospital (Other)
Collaborators: AC Immune SA (Industry)
Responsible Party: Principal Investigator, Oskar Hansson, Professor, Skane University Hospital
Other Study IDs: A-synuclein-PET-study
Record Dates: First submitted 2021-09-23; First posted 2021-10-05 (Actual); Last update posted 2021-10-05 (Actual); Status verified 2021-09

CONDITIONS: Parkinson Disease; Dementia With Lewy Bodies; Multiple System Atrophy; Corticobasal Degeneration; Progressive Supranuclear Palsy
MeSH Terms: conditions — Parkinson Disease; Lewy Body Disease; Multiple System Atrophy; Corticobasal Degeneration; Supranuclear Palsy, Progressive

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (6):
- Parkinson's Disease: Patients with Parkinson's Disease. Patients will undergo [18F]ACI-3847 PET, [18F]DOPA PET and MRI. Up to 20 patients will be scanned
- Dementia with Lewy Bodies: Patients with Dementia with Lewy Bodies. Patients will undergo [18F]ACI-3847 PET, [18F]DOPA PET and MRI. Up to 10 patients will be scanned
- Multiple System Atrophy: Patients with Multiple System Atrophy. Patients will undergo [18F]ACI-3847 PET, [18F]DOPA PET and MRI. Up to 10 patients will be scanned
- Corticobasal Syndrome: Patients with Corticobasal Syndrome. Patients will undergo [18F]ACI-3847 PET, [18F]DOPA PET and MRI. Up to 10 patients will be scanned
- Progressive Supranuclear Palsy: Patients with Progressive Supranuclear Palsy. Patients will undergo [18F]ACI-3847 PET, [18F]DOPA PET and MRI. Up to 10 patients will be scanned
- Healthy controls: Healthy contols. Contols will undergo [18F]ACI-3847 PET, [18F]DOPA PET and MRI. Up to 20 patients will be scanned

SUMMARY:
The aim of the project is to develop the first alpha-synuclein (a-syn)-specific PET tracer. The research phase will exploit ACI's proprietary MorphomerTM library and extensively optimized screening workflow.

Promising PET-tracer candidates will be tested for their ability in detecting a-syn pathology in patients with a range of Parkinsonian conditions with different a-syn levels and distributions, comprising hereditary forms of PD and other synucleinopathies.

DETAILED DESCRIPTION:
Aims:

Today there is no way of detecting a-synuclein pathology in life, and thus the diagnoses of Parkinson's Disease (PD) and the closely related synucleinopathies Dementia with Lewy Bodies (DLB) and Multiple system atrophy (MSA) are clinical diagnoses, that can be supported by dopamine (F-DOPA) imaging and biomarkers (f.ex cerebrospinal fluid neurofilament light chain), but where the ultimate diagnosis is not certain until at post mortem investigation of the brain.

The general aim of this study is to assess a newly developed positron emission tomography (PET) tracers for a-synuclein and to study the ability of the tracer in detecting the underlying pathology in PD, DLB and MSA. If the PET tracers can detect the pathology reliably our hope is that this tracers can assist in future clinical trials for PD, DLB and MSA.

Primary aim

• to assess the brain a-synuclein load in vivo using [18F]ACI-3847 PET in MSA, DLB and Parkinson's disease

Secondary aims

* to explore the correlation in these patients between a-synuclein load assessed by [18F]ACI-3847 PET and clinical features including cognitive impairment and severity of neurological symptoms
* to detect a-synuclein pathology assessed by [18F]ACI-3847 PET in Parkinson cases with a duplication in the gene coding for a-synuclein

Background:

Clinical presentation: Neurodegenerative disorders mainly affect the elderly population and approximately 1% of the population above 60 are affected by PD. DLB is likely underdiagnosed, but represent approximately 10% of the patients in a specialist dementia center setting. MSA is more uncommon and is often mistaken for PD, but carries a much worse prognosis. Due to the poor prognosis of MSA it is important to as early as possible be able to give a correct diagnosis.

The diagnoses of PD, DLB and MSA are today mainly clinical diagnoses. The diagnosis of PD is based on the triad of symptoms: rigidity, resting tremor and bradykinesia of movement, followed by a rapid and sustained response of symptoms to levodopa treatment. Further, the loss of dopaminergic neurons can be visualized with PET-imaging of dopamine storage capacity (18F-DOPA PET). At symptom onset of PD it has been estimated that 50-70% of dopaminergic cells are already lost, making it more difficult to successfully treat the disease to halt or slow down disease progression. MSA causes similar symptoms as PD, and is often mistaken for PD, but patients gradually also develop autonomic failure, with varying heart rate and blodpressure, causing falls due to ortostatic drops in blood pressure. F-DOPA PET again shows a loss of dopaminergic cells in the midbrain, but the levodopa response is much attenuated in MSA. DLB shows similar symptoms of bradykinesia and rigidity, but also early on changes in cognition and visual hallucinations.

Neuropathology: PD, DLB and MSA are all caused by aggregation of a-synuclein in the brain. The midbrain and the brainstem is first affected in PD, and later in the disease the pathology spreads throughout the neocortex. In DLB the a-synuclein often also involves the occipital neocortex and limbic brain structures in addition to the midbrain. In MSA the pathology affects the brain stem and basal ganglia, but also often the cerebellum.

Diagnostic work-up: As stated earlier there is today no reliable way to verify the diagnoses or the a-synuclein in life. In this study we will include also 18F-DOPA PET that is today the state-of-the-art technique for detecting a loss of dopamine producing cells in the midbrain. 18F-DOPA PET will strengthen the diagnostic accuracy, but there are still pitfalls even when using 18F-DOPA PET for diagnosis. For example the Parkinson-related disorders Progressive Supranuclear Palsy (PSP) and Corticobasal Degeneration (CDB), that both show dopamine cell loss and a decreased 18F-DOPA retention in addition to PD-like symptoms like bradykinesia and rigidity, but that both are caused by tau pathology and not a-synuclein pathology. It is well known that the diagnostic accuracy of some of the diagnoses with parkinsonism is at best moderate and that many diagnoses will have to be corrected at autopsy.

Our hope is that [18F]ACI-3847 PET in the long run will help in the differential diagnosis against PSP and CBD, but also that the different patterns of a-synuclein accumulation in PD, DLB and MSA will provide a useful tool in tracking disease progression within the synucleinopathies.

Treatment trials: There are currently no treatments that slow down or stop PD, DLB or MSA. There are large efforts to develop therapies (e.g. immunotherapies) that remove aggregated a-synuclein from the brains of the affected patients. However, there is no methods available today that can be used to study whether such treatments really affect the levels of abnormal a-synuclein in the living human brain. If [18F]ACI-3847 PET can visualize the a-synuclein aggregates, then it might be used in the future to evaluate whether novel therapies can remove a-synuclein from the brain of living humans.

Participants:

Patients with PD, DLB, MSA, PSP and CBD and Healthy controls.

Inclusion criteria - patients

* Age 50-100 years.
* Fulfill the criteria for PD, DLB, MSA, PSP or CBS.
* Speaks and understands Swedish to the extent that an interpreter was not necessary for the patient to fully understand the study information and cognitive tests.

Exclusion criteria - patients

* Significant unstable systemic illness or organ failure, such as terminal cancer, that makes it difficult to participate in the study.
* Current significant alcohol or substance misuse.
* Refusing MRI or PET.

Inclusion criteria - healthy controls

* Age 50-100 years
* Absence of cognitive symptoms or parkinsonism as assessed by a physician with special interest in cognitive disorders.
* Speaks and understands Swedish to the extent that an interpreter is not necessary for the patient to fully understand the study information and cognitive tests.

Exclusion criteria - healthy controls

* Significant unstable systemic illness or organ failure, such as terminal cancer, that makes it difficult to participate in the study.
* No significant neurological or psychiatric disease.
* Current significant alcohol or substance misuse.
* Refusing MRI or PET.

Methods:

Positron Emission Tomography [18F]ACI-3847 PET (a-synuclein PET) will be performed in all participants. 185 MBq (5 mCi) [18F]ACI-3847 is injected intravenously via an intravenous cathether. Data acquisition is started at the time of injection and continues over 100 minutes (0-100 min). During this time the patient will need to keep as still as possible. Image data will be collected on GE Discovery MI PET/CT cameras as LIST mode data (raw data) and be reconstructed after acquisition and attenuation correction. Arterial sampling will be performed in a subset of individuals.

[18F]DOPA PET for assessment of remaining dopamine producing cells will be performed by intravenous injection of 185 MBq (5 mCi) [18F]DOPA. Data acquisition is started at either at the time of injection and continues over 110 minutes, or starts 90 min after injection and continues for 20 minutes. No arterial blood sampling is needed for this scan.

Magnetic Resonance Imaging 3 Tesla MRI (Siemens Prisma) will be done in all participants. No contrast-enhancing agent will be used.

ELIGIBILITY:
Inclusion Criteria:

* Age 50-100 years.
* Fulfill the criteria for PD, DLB, MSA, PSP or CBS. Alongside with these participants patients with duplications in the gene coding for a-synuclein will be included.
* Absence of cognitive symptoms or parkinsonism as assessed by a physician with special interest in cognitive disorders (Healthy controls).
* Speaks and understands Swedish to the extent that an interpreter was not necessary for the patient to fully understand the study information and cognitive tests.

Exclusion Criteria:

* Significant unstable systemic illness or organ failure, such as terminal cancer, that makes it difficult to participate in the study.
* Current significant alcohol or substance misuse.
* Refusing MRI or PET.

Min Age: 50 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Study Population: Patients with synucleinopathies (PD, DLB and MSA), patients with other Parkinson Plus disorders (CBS, PSP) and controls.
Sampling Method: Non-Probability Sample
Enrollment: 12 (Actual)
Dates: Start 2021-07-15 (Actual); Primary Completion 2021-09-01 (Actual); Study Completion 2021-09-01 (Actual)

PRIMARY OUTCOMES:
Detection of alpha-synuclein pathology | July 2020 - August 2022
  Assess the ability of alpha-synuclein tau tracer [18F]-ACI3847 in detecting tau pathology in synucleinopathies.

CONTACTS AND LOCATIONS:
Overall Officials: Oskar Hansson, Professor, Principal Investigator — Skane University Hospital
Locations (1):
- Skåne University Hospital, Dept of Neurology, Lund, Skåne County, Sweden

IPD SHARING:
Plan to Share IPD: Undecided